CLINICAL TRIAL: NCT06472518
Title: Prospective Randomised Multicentre Medico-economic Evaluation of Pharmaco Mechanical Thrombolysis Associated With Anticoagulation Compared With Anticoagulation in the Acute Phase of Very Symptomatic Proximal Venous Thrombosis of the Lower Limbs.
Brief Title: Pharmaco Mechanical Thrombolysis Associated With Anticoagulation Compared With Anticoagulation in the Acute Phase of Very Symptomatic Proximal Venous Thrombosis of the Lower Limbs.
Acronym: PMT-DVT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC22_0472
Record Dates: First submitted 2024-04-02; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Iliofemoral Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pharmaco mechanical thrombolysis (Experimental): thrombolysis intervention combined with anticoagulant treatment with direct oral anticoagulants
  Interventions: Device: pharmaco mechanical thrombolysis
- oral anticoagulant alone (Active Comparator): a reference treatment arm for patients receiving direct oral anticoagulant alone and stenting angioplasty in case of venous claudication or moderate post-thrombotic syndrome six months after the initial thrombosis.
  Interventions: Device: pharmaco mechanical thrombolysis

INTERVENTIONS:
Device: pharmaco mechanical thrombolysis — arm with the pharmaco mechanical thrombolysis intervention combined with anticoagulant treatment with direct oral anticoagulants

SUMMARY:
* Iliofemoral DVTs (IF DVTs) are vascular disorders associated with high morbidity and mortality, which can be complicated by long-term post-thrombotic syndrome (PTS).
* Pharmaco mechanical thrombolysis (PMT) is an innovative endovascular technique involving in situ fibrinolysis of the thrombus in the acute phase of thrombosis, followed by mechanical extraction by fragmenting the thrombus.
* The American ATTRACT study showed that management by catheter-directed thrombolysis and/or PMT in the acute phase is safe and effective at 2 years in a subgroup of DVTif compared with anticoagulation (18% moderate or severe SPT with thrombolysis vs. 28% without thrombolysis).
* PMT-DVT will be the first study to assess the medium (30 months) and long-term (60 months) efficacy of PMT in the French context, using data from the French National Health Data System.

DETAILED DESCRIPTION:
Patients with acute iliofemoral thrombosis will be included in the study after consent. They will be randomized to pharmaco-mechanical thrombolysis combined with anticoagulant therapy with direct oral anticoagulant versus direct anticoagulant therapy alone. They will be monitored, and patients in the anticoagulation-only group may undergo stenting angioplasty in the chronic phase if they present a moderate post-thrombotic syndrome or venous claudication. At the end of 30 months, a medico-economic analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agreed to participate in the study and gave oral consent.
* Patient affiliated to a social security scheme
* Iliac and/or common femoral venous thrombosis
* Recent thrombosis less than or equal to 14 days since qualifying imaging or less than or equal to 21 days since onset of symptoms

And at least 1 of the following criteria:

* Visual analog scale greater than or equal to 5 and/or
* Venous claudication and/or
* Increase in thigh circumference greater than or equal to 5% compared with contralateral thigh.

Exclusion Criteria:

* Patients with superficial femoral or popliteal venous thrombosis without involvement of the common femoral or iliac veins.
* Patients with isolated thrombosis of the inferior vena cava, without extension to the iliac veins.
* Thrombosis of inferior vena cava proximal to the renal veins.
* Minors, pregnant women, adults under guardianship.
* Chronic renal failure with creatinine clearance below 30ml/min according to Cockroft.
* Ischaemic phlebitis: proximal venous thrombosis associated with limb ischemia and impaired arterial flow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Cost-utility analysis | 30 month
  Cost-utility analysis of the economic efficiency of the PMT strategy compared with the anticoagulation strategy for the treatment of DVT from a collective perspective and a 30-month time horizon

SECONDARY OUTCOMES:
Number of patients with Villalta score greater than or equal to 10 | 30 month
  Number of patients with Villalta score greater than or equal to 10
Number of patients with Villalta score greater than or equal to 15, or presence of ulceration | 30 month
  Number of patients with Villalta score greater than or equal to 15, or presence of ulceration
Number of major hemorrhages and number of clinically relevant non-major hemorrhages according to ISTH criteria | 1, 30 and 60 month
  Number of major hemorrhages and number of clinically relevant non-major hemorrhages according to ISTH criteria
Number of patients with pain greater than or equal to 7 as assessed by the visual analog scale, or the presence of venous claudication, or lower-limb edema with a circumference greater than 20% of the contralateral leg, or failure to return to work. | 1 month
  Number of patients with pain greater than or equal to 7 as assessed by the visual analog scale, or the presence of venous claudication, or lower-limb edema with a circumference greater than 20% of the contralateral leg, or failure to return to work.
VEIN-QOL | 1,30 and 60 month
  overall assessment by questionnaire
CIVIQ 20 | 1,30 and 60 month
  score 0 to 100
SF36 scores | 1,30 and 60 month
  score 0 to 100
Number of patients with onset of venous claudication | 30 month
  Number of patients with onset of venous claudication
Number of patients with a trophic disorder, assessed by clinical examination | 60 month
  Number of patients with a trophic disorder, assessed by clinical examination
Incremental cost-utility ratio of MPT compared with anticoagulation strategy | 60 month
  Incremental cost-utility ratio of MPT compared with anticoagulation strategy
Net financial impact over 5 years of TPM distribution | 60 month
  Net financial impact over 5 years of TPM distribution

IPD SHARING:
Plan to Share IPD: No